

## SIVAS CUMHURIYET ÉNIVERSITESI GIRIŞIMSEL OLMAYAN KUNİK ARAŞTIRMALAR ETİK KURULU KARAR FORMU

ARASTRONANIN ACIK ADI

Ober Oswokul Öğrencilerinik Sağlığı Golqtirme Modeline Dayalı Verilen Planh Eginnum Yaşının Sulli Davramşları ve Kilin Yönesimine Edkini

| | Belge Adv | | Taribi | Versiyon<br>Numerasi | | DIII | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| dias. | AKASSTRMA P | имскови | | | Dido | () [S]. | Trigit | ine E | 18 | MA. |
| PRÉCEDE ENDREELEN<br>MELGELEN | 00.000.050000 | ифолоти счоту го | 999 | | fud | <b>Ø</b> | | un 🗆 | | e CI |
| | DESCRIPTIONS | | | | Tark | | | m D | - UD | e C |
| | | Hoter Mile | | | === | - 69 | Alatin | | | |
| | ANASTROOPS | PROBLEM . | - 10 | | | | | | | |
| | SOME RUN R | | 0 | | | | | | | _ |
| | DATER | | - D | | - | | | - | _ | - |
| KARAK | Kerne Ser 2844 | 8110 | 1 Table 11/00/00 | Table 0.00.002 | | | | | | |
| rbs secret | LIP CALISS | Library Arms | AYAN MEDIN ARA<br>peralir Hakkinda Yos<br>(Coverales) Girginia | estruction Del State | ALL YES | director | Kara | rest. Hell | Hada Na | dapen |
| USKANTI | CNVANT/ADD | | iller Yoldman | | | Tall Little | 2000 | | | |
| Larranchide Segreta | | Lineshi Niss | Karumi | Ela | Linese | | Advationing IIII<br>Stale | | Kittine - | |
| | 36les | has harde yo this. | Strain Combination Com-<br>Try Flamburs | - 1 D | K 33 | 11 | 1100 | e m | ΝП | 1111 |
| haven)<br>of D. Hous | ar Bragato | her hards ye bid. Discharge to Discond. | | THAM. VIT | K 53<br>K 50 | Esta. | 700 | 6 E | 10 | In. |
| licanen)<br>inc. Dr. Hows<br>linghan Yard<br>and Dr. House | or Diagno<br>omices)<br>car Applies | MARKET SE | Try Function Seven Calebrary In Chin | man. r.D | 160 | e Er | 1100 | HH | CONTROL OF | TA JIA |
| liganes)<br>ing Di Hjeen<br>leghan Yard<br>and Di Hanes<br>Augustila) | ar Bugos<br>umorni<br>nan Avidan | Bulanes is Deciral | Top Flantifice: Reven C undustryer Over Jugodi Tutter und Festige Proge Comburrors Dated | men rB | k.83 | € E3 | #Ø | 68 | #0 | |
| House, Dr. House<br>Hephan Varia<br>and Dr. House<br>Magnetile; | or Rugos<br>venore)<br>sur Avidan<br>(Karber) | Sections to Decemb<br>Light Sections<br>Exhaulter to | Top Functions forms Charlestyn Liter legisk form un Fonde frequ Charlestyn Char fog Fakalture frezo Charlestyn Char fogfak fokalter Fokula litina Chiralestyn Fokula Dog Fakaltig Fokula | entale FD | 4.53<br>4.D | : EI | #8<br>#8 | · 8 | 10 | MAN T |
| House, D. House<br>Replace Varia-<br>and Dr. House<br>Kapacalleri<br>and The Moura<br>Lot the House<br>Lot the House | or Bugos<br>sensors)<br>sur Aviden<br>(Surtes)<br>or Donne | Tricks for examina Fight Supplies for Historical Displacements Francis Displacements Assessed | Top Families Server Construction Livery Legisla Terres on Linear Server Construction Construction Server Construction Construction Server Construction Construction Day Education Federal Server Construction Constr | enter ES | 4 (S)<br>4 (D)<br>4 (S) | : D<br>: D<br>: D | #8<br>#8<br>#8 | 6 13<br>6 13 | 0.00 | MAN TO |
| House, Dr. House<br>Hephan Varia<br>and On House<br>Magnerile;<br>and He More<br>for the Mary<br>Tot the Hand | or Rugos<br>veneral<br>par Nodas<br>(Sarbei)<br>pr Dones | Suctions to Decemb<br>Links Scroburns<br>Fish Sugligator<br>Hateshiller Homosolip<br>Expens Dig Steeres | Top Function forms Charlestyn Liter legisk formum Funch form Charlestyn Char fog Fulcifum form Charlestyn Char fog Fulcifum form Charlestyn Char fog Fulcifum form Charlestyn Char fog Fulcifum form Charlestyn Char fog Fulcifum formum Charlestyn Char fog Fulcifum formum Charlestyn Char fog Fulcifum formum Charlestyn Char fog Fulcifum formum Charlestyn Char formum Charlestyn Charles | entale FD street FD cores, FD cores, FD cores, FD | 4 (S)<br>4 (D)<br>4 (S) | 10 | #8<br>#8<br>#8 | 6 13<br>6 13 | | |
| Horneys Heyber Vers Heyber Vers Heyber Vers Hagerrile Hof De Horn Jos De Han Jos De | or Rugos<br>veneral<br>par Nodas<br>(Sarbei)<br>pr Dones | Total Secretaria Talka Secretaria Esch Suglige Se Historial Dep Section Assure Factorial | Top Families Server C wellscript Cree Jagod Town on T solds Server C wellscript Cree Top Fakisher Server C wellscript Cree Dop Fakisher Dop Fakisher Server C wellscript Cree Top Fakisher Server C wellscript Cree Top Fakisher Server C wellscript Cree Top Fakisher Server C wellscript Cree Top Fakisher Server C wellscript Cree Top Fakisher Server C wellscript Cree Server C wellscript C wel | TOTAL FOR | 4 (S)<br>4 (D)<br>4 (D)<br>4 (D) | 0 0 0 | 11 (S)<br>11 (S)<br>11 (S)<br>11 (S)<br>11 (S) | 6 8<br>6 8<br>6 8<br>6 8<br>8 | 0 0 0 | |
| | or Dago<br>season)<br>ser Ayden<br>(Kathali<br>or Done)<br>ling | Total Services Total Services Fixe Supliquire Historialist Throughout Experia Dig State or Assessive Experialist Exp | Top Familians Beyon C unduring in Copy Ingles To the con- I make to the Top TableStorm Server C unduring the Copy Industry Copy Industrial Top TableStorm Dog I demanding TableStorm Copy Industrial TableStorm Server Cumburger Copy Top Endosters Server Copy Top Endosters Server Cumburger Copy Top Endos | TOTAL FOR | 4.50<br>4.50<br>4.00<br>4.00<br>4.00 | | #80<br>#80<br>#80<br>#80<br>#80 | 6 (E)<br>6 (E)<br>6 (E)<br>8 (E)<br>8 (E) | | |
| transmitted to the second of the state of th | or Rugos<br>sensoral<br>car Avolen<br>Charteet<br>or Doma<br>regulatery<br>sensoral Alice<br>Abrest Alice<br>Fine German | Distance of Decemb<br>Light Services<br>Expending or<br>Haladeller Homorely<br>Expend Dig Salacon<br>Assesse<br>Factorists<br>(Services) | Top Familians Service Conduction Congression Congression Conduction Conduction Congression Congressio | ement E E E E E E E E E E E E E E E E E E E | 40<br>40<br>40<br>40<br>40 | 10 10 10 10 | # 20 m 20 m 20 m 20 m 20 m 20 m 20 m 20 | 6 28 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | | |

A STATE OF

His Kumi Başkamı Unvim/Adi/Seyath Prof. Br Obley Vidermi limea.



## SIVAS CUMBILIRIVET (INIVERSITES) UBUSIANSEL OLMAYAN KLINİK ARAŞTIRMALAR ETİK KURULU KARAR FORMU

ARASTIBNIANIN ACTICADI

Obez Ortnokul Öğrencüerinde Sağlağı Geleştirme Modeline Dayalı Vertien Planti Egimuin Yugam Stills Davranglari ve Kilin Vonetimine Efkini

ULUSA.

STREET, MAKEUR D

coulurs cord

| (7) | ETIK KURULUN ADI | Contractor Conversion Girsginnet Olmayon Klimic Aragormatur<br>Karpilo<br>Saves Comburiyar Oniversion Up Febilioni Dekantigo,<br>Tap Taribi ve Paik Anabilim Dali<br>TR-58140 Merker Saves |
|---|---|---|
| BESCHERU<br>BESCHERU | AÇIK ADRESÎ. | |
| 3 | TELEFON | 0.346 487 20.92 |
| | EAKS<br>E-PONEA | gotack2014@spnail.com |
| п они кум | SECREPANCE SORDMENT ARASTONACI<br>LWANDARDSOYADI | Dr. Ogr. Cycat Senna Ziolic |
| | ROOMERY CONTROL OF A STANISH ALANI | Halk Soglige Hemsireligi |
| | ACASTINGGENN HULLINDOĞU<br>MÜRKEM | Sives Combanyot Üniversitesi Saglik Bilimlen Faktisesi<br>Hempirelik Bölüsü, Halk Sagligi Bempireliği Azabilin Dalı |
| = | DESTERLEYED | |

Delitora lezi

DESCRIPTIONS

Bulk Kurul Baskass

University Ada/Seyndr, Prof. Dr. Cintay Yildmin.

DESTRUEPHENDLY ASAL TONNECET

AUCKS TOURIAMOST TÜRCT.

ARABIBUAYA KATILAS MERKEZLER

ferres: